CLINICAL TRIAL: NCT05286710
Title: Clinical Study On The Improvement Of Rheolytic Thrombectomy For Acute Deep Vein Thrombosis Of Whole Lower Limb By Primary Popliteal Vein Thrombosis Clearance
Brief Title: Rheolytic Thrombectomy For Acute Deep Vein Thrombosis Of Whole Lower Limb
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: First People's Hospital of Hangzhou (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Affiliated Hospital of Nantong University (Other); Chengdu University of Traditional Chinese Medicine (Other); Second Affiliated Hospital of Suzhou University (Other); Liuzhou Workers' Hospital (Other Government); Shanghai Pudong New Area People's Hospital (Other); Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The Reformation Study
Record Dates: First submitted 2022-03-06; First posted 2022-03-18 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Deep Vein Thrombosis
Keywords: pharmacomechanical thrombectomy
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified access group (Experimental): modified access: PMT was performed via distal calf venous access or contralateral femoral access
  Interventions: Device: pharmacomechanical thrombectomy (PMT)
- traditional access group (Active Comparator): traditional access: PMT was performed via ipsilateral popliteal venous access
  Interventions: Device: pharmacomechanical thrombectomy (PMT)

INTERVENTIONS:
Device: pharmacomechanical thrombectomy (PMT) — After randomization patients will be allocated to pharmacomechanical thrombectomy (PMT) via ipsilateral popliteal venous approach or to PMT via distal calf venous approach, bail-out contralateral femoral access can be used if puncture was failed in calf vein. After PMT treatment, residual thrombus was reevaluated by ascending venography. Catheter-directed thrombolysis (CDT) was conducted if there was residual thrombus. Stenosis of iliac vein was assessed by multiangle venography and intravascular ultrasound (IVUS) was used if necessary. Percutaneous balloon angioplasty (PTA) was conducted if there was >50% stenosis of the diameter of the iliac vein. A stent was placed if the residual stenosis was >50% after PTA treatment.

SUMMARY:
Ipsilateral popliteal venous the most common access for pharmacomechanical thrombectomy (PMT) in the treatment of acute deep venous thrombosis (DVT), but the result was not satisfactory. The investigators adjust the access to improve the thrombus clearance rate and reduce the incidence of post-thrombotic syndrome (PTS).

DETAILED DESCRIPTION:
Acute deep venous thrombosis (DVT) with whole lower limb involved is associated with significant post thrombotic morbidity. Both of deep venous occlusion and valvar reflux increase the risk for development of post-thrombotic syndrome (PTS). Early removal of iliofemoral thrombosis by pharmacomechanical thrombectomy (PMT) may reduce the incidence of PTS. In general, ipsilateral popliteal venous the most common access for PMT. However, from this approach, it's hard to remove the thrombosis in the distal popliteal vein. So, the investigators hypothesize that the residual thrombus and slow blood-flow in the in-flow may weakened the efficacy of PMT, and by adjusting vein access approach could improve the thrombus clearance rate and reduce the incidence of PTS for whole leg DVT.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years old;
* Acute DVT with clinical symptoms occurred less than 14 days since the onset of disease;
* DVT with thrombosis involving the iliac vein, common femoral vein, distal popliteal vein, and/or calf vein;
* Informed consent signed by patients.

Exclusion Criteria:

* Patients with the previous history of the same side of lower-limb DVT;
* Patients with plasma Creatinine level greater than 180umol/L;
* Patients who are contraindicated to thrombolysis;
* Patients with inferior vena cava thrombosis;
* Patients who are known to be allergic to heparin, low molecular weight heparin, or contrast agent;
* Patients who have participated in a clinical trial in the past three months;
* Women during pregnancy and lactation
* Patients with other diseases that may cause difficulty in the study or significantly shorten the life expectancy of patients (<2 years);
* Patients with autoimmune thrombopathy or thrombocytopenia (platelets < 80·10⁹/L);
* Patients who are unable or unwilling to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-thrombotic syndrome (PTS) | 24 months
  Incidence of post-thrombotic syndrome (PTS) at post-interventional 24 months

SECONDARY OUTCOMES:
Immediate patency rate | immediately after lonely mechanical thrombectomy
  Percentage of patency rate immediately after lonely mechanical thrombectomy
Total time of interventional surgery | immediately after interventional surgery
  Total time measured by hours of interventional surgery (Including duration of subsequent catheter directed thrombolysis)
Total dosage of urokinase | immediately after interventional surgery
  Total dosage measured by units of urokinase used for procedure
Patency rate of lower limb vein | post-interventional 12 and 24 months
  Percentage of patency rate of lower limb vein at post-interventional 12 and 24 months
Deep venous valve function evaluation | post-interventional 12 and 24 months
  Deep venous valve function evaluation by ultrasound at post-interventional 12 and 24 months
Quality of life evaluated by 36-Item Short Form Health Survey (SF-36) | post-interventional 3, 6, 12 and 24 months
  Quality of life evaluated by 36-Item Short Form Health Survey (SF-36). The change in SF-36 Physical and Mental Component Scales from baseline to 24 months will be compared between the two groups using a t-test. A difference of 5 points on each scale is considered to be clinically relevant. In addition, a linear mixed model analysis of the repeated assessments (3, 6, 12, and 24 months) with baseline scores as a covariate will be used to investigate the changes over time, and if they differ by treatment arm.
Venous Insufficiency Epidemiological and Economic Study Quality of Life (VEINES-QOL) score | post-interventional 3, 6, 12 and 24 months
  Venous Insufficiency Epidemiological and Economic Study Quality of Life (VEINES-QOL) score at post-interventional 24 months; The minimum value is 21, and the maximum value is 118. The higher scores mean a better outcome.
European quality of life 5-dimension 5-level (EQ-5D-5L) score | post-interventional 3, 6, 12 and 24 months
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Re-intervention rate | within 24 months after operation
  Percentage of re-intervention rate within 24 months after operation
Rate of catheter-directed thrombolysis | immediately after interventional surgery
  Percentage of catheter-directed thrombolysis after mechanical thrombectomy

OTHER OUTCOMES:
Safety outcomes - procedural complications | Within 30 days after intervention
  Procedural complications such as hematoma at the puncture site, hemoglobinuria or hemolytic jaundice
Safety outcomes - major bleeding events | Within 24 months after intervention
  Major bleeding events according to the International Society on Thrombosis and Haemostasis (ISTH)
all-cause death | Within 24 months after intervention
  All-cause death during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ye, M.D., Study Director — Department of Vascular Surgery, Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ni Q, Ye X, He C, Zhao H, Lou W, Zhuang H, Sang H, Wu Z, Ye M. Improvement of rheolytic thrombectomy for acute deep vein thrombosis of the whole lower limb by primary popliteal vein thrombosis clearance: protocol for a prospective, multicenter, randomized controlled trial (the Reformation study). BMJ Open. 2025 Jun 3;15(6):e089797. doi: 10.1136/bmjopen-2024-089797. PMID 40461147